CLINICAL TRIAL: NCT05420129
Title: Side Effects of the Use of the Mandibular Advancement Device for Treatment of Obstructive Sleep Apnea on Dental Occlusion and Masticatory Function
Brief Title: Side Effects of the Mandibular Advancement Device for Apnea Treatment on Dental Occlusion and Masticatory Function
Status: Withdrawn | Type: Observational
Why Stopped: The researcher who would recruit the participants is not longer available
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor, University of Barcelona
Other Study IDs: HOUB2021/039
Record Dates: First submitted 2022-05-24; First posted 2022-06-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MAD. Mandibular advancement Device: Patients diagnosed with Obstructive Sleep Apnea and treated with MAD
  Interventions: Device: MAD Therapy
- CPAP. Continuous Possitive Airway Pressure: Patients diagnosed with Obstructive Sleep Apnea and treated with CPAP
  Interventions: Device: CPAP Therapy

INTERVENTIONS:
Device: MAD Therapy — Participants will be treated with a Mandibular Advancement Device therapy
  Groups: MAD. Mandibular advancement Device
Device: CPAP Therapy — Participants will be treated with a Continuous Positive Airway Pressure therapy
  Groups: CPAP. Continuous Possitive Airway Pressure

SUMMARY:
This study evaluates the effect of the use of mandibular advancement devices (MAD) on dental occlusion and masticatory function during the first two years of obstructive sleep apnea (OSA) treatment.

52 participants diagnosed with obstructive sleep apnea will be studied, 26 will be treated with MAD and 26 participants will be treated with continuous positive airway pressure (CPAP) as a control group.

Participants will perform masticatory tests to assess masticatory performance in comminute and mixing capacity. Masticatory satisfaction perceived by the participants will be evaluated by questionnaires. Occlusal contact area and other occlusal characteristics will be assessed using occlusal silicone and T-Scan registrations and 3D digital models obtained with intraoral scan. Data collection will be performed before treatment with MAD or CPAP, and at 3, 6, 12, and 24 months from the start of treatment.

DETAILED DESCRIPTION:
This prospective observational non-randomized clinical study aims to assess the effect of use MAD on masticatory performance. 52 subjects diagnosed with OSA will participate in this study divided into two different groups: 26 treated with MAD and 26 treated with CPAP. Data collection will be carried out before the start of treatment of the two modalities and at 3, 6, 12 and 24 months after starting the treatment. The intervention of the study will be based on execute chewing tests to evaluate masticatory performance from artificial food. Other aspects of matsticatory function would be also explored like subjective masticatory performance and jaw function limitation, dental position and occlusion, bite force or dental mobility. Artificial food tests will evaluate masticatory performance in comminute and mixing ability to determine the degree of reduction in masticatory performance produced by the use of MAD after 3 months of treatment. The main variable to be studied will be the median particle size of silicone tablets from Optozeta's test. This test is based on chewing 2 grams of silicone tablets inside a latex bag in order to evaluate their degree of comminution. The greater of grinded silicone, the greater of chewing performance. Another masticatory performance test will also be carried out is evaluation subject's mixing capacity with a two-colour chewing gum test. Degree of mixing of two colours of the gum will be checked after 40 chewing cycles. The more uniformity of the colour obtained, the more mixing ability the subject will demonstrate. A CPAP group control will be used, which will additionally allows us to know if this treatment has effects on dental position, occlusion and masticatory performance.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with OSA by polisomnography (IAH>15).

Exclusion Criteria:

* Be treated with MAD or CPAP during more than 3 months in the lasts 5 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sleep apnea and treated with CPAP or MAD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in masticatory perfomance at 6 months | Before treatment and 6 months after treatment
  The masticatory performance will be evaluated by assessing the degree of comminution of the silicon test food (Median particle size). The particles from five trials (10 g) will be dried and passed through a series of eight sieves (0.25, 0.425, 0.85, 2, 2.8, 3.15, 4, and 5.6 mm) while being shaken for 6 min. Once the cumulative weight distribution of the sieve contents will be determined, the median particle size (MPS) will be calculated for each subject using the Rosin-Rammler equation [Qw (X) = 1 - 2E-(X/ X50)b], where Qw (X) is the fraction of particles by weight with a diameter smaller than X; X50 (or MPS) is the size of a theoretical sieve through which 50% of the weight would pass; and b describes the breadth of the particle size distribution. Therefore, the lower the MPS, the better the masticatory performance. Participants will perform masticatory tests before and 6 months after treatment.
Change in masticatory perfomance at 24 months | Before treatment and 24 months after treatment
  The masticatory performance will be evaluated by assessing the degree of comminution of the silicon test food (Median particle size). The particles from five trials (10 g) will be dried and passed through a series of eight sieves (0.25, 0.425, 0.85, 2, 2.8, 3.15, 4, and 5.6 mm) while being shaken for 6 min. Once the cumulative weight distribution of the sieve contents will be determined, the median particle size (MPS) will be calculated for each subject using the Rosin-Rammler equation [Qw (X) = 1 - 2E-(X/ X50)b], where Qw (X) is the fraction of particles by weight with a diameter smaller than X; X50 (or MPS) is the size of a theoretical sieve through which 50% of the weight would pass; and b describes the breadth of the particle size distribution. Therefore, the lower the MPS, the better the masticatory performance. Participants will perform masticatory tests before and 24 months after treatment.

SECONDARY OUTCOMES:
Change in masticatory mixing ability at 6 months | Before treatment and 6 months after treatment
  Masticatory mixing ability will be measured using the standard deviation of red channel in RGB image of a colour histogram. It will be assessed by doing a two-colour gum chewing test. Higher values of the standard deviation of red channel will indicate poor masticatory mixing ability. Participants will perform masticatory tests before and 6 months after treatment.
Change in masticatory mixing ability at 24 months | Before treatment and 24 months after treatment
  Masticatory mixing ability will be measured using the standard deviation of red channel in RGB image of a colour histogram. It will be assessed by doing a two-colour gum chewing test. Higher values of the standard deviation of red channel will indicate poor masticatory mixing ability. Participants will perform masticatory tests before and 24 months after treatment.
Change in the degree of satisfaction in masticatory function at 6 months | Before treatment and 6 months after treatment
  The change in the degree of satisfaction in masticatory function at 6 months will be assessed by asking the question "How satisfied are the participants with their masticatory function? using a 0-10 point scale, considering 0 totally dissatisfied and 10 totally satisfied. Participants will rate before treatment and 6 months after treatment.
Change in the degree of satisfaction in masticatory function at 24 months | Before treatment and 24 months after treatment
  The change in the degree of satisfaction in masticatory function at 24 months will be assessed by asking the question "How satisfied are the participants with their masticatory function? using a 0-10 point scale, considering 0 totally dissatisfied and 10 totally satisfied. Participants will rate before treatment and 24 months after treatment.
Change in chewing ability at 6 months | Before treatment and 6 months after treatment
  The change in chewing ability will be assessed by filling out a questionnaire about differents types of food. For each food, the participant will ask the question "How able are the participants to chew this food? using a 0-10 point scale, considering 0 totally unable and 10 totally able. Participants will rate before treatment and 6 months after treatment.
Change in chewing ability at 24 months | Before treatment and 24 months after treatment
  The change in chewing ability will be assessed by filling out a questionnaire about differents types of food. For each food, the participant will ask the question "How able are the participants to chew this food? using a 0-10 point scale, considering 0 totally unable and 10 totally able. Participants will rate before treatment and 24 months after treatment.
Change in jaw functional limitation.at 6 months | Before treatment and 6 months after treatment
  The change in jaw functional limitation will be assessed by filling out the Jaw Functional Limitation Scale (JFLS-20), with the question: "For each of the items, indicate the level of limitation anbout the following functions", using a 0-10 point scale, considering 0 no limitation and 10 severe limitation. Participants will rate before treatment and 6 months after treatment.
Change in jaw functional limitation.at 24 months | Before treatment and 24 months after treatment
  The change in jaw functional limitation will be assessed by filling out the Jaw Functional Limitation Scale (JFLS-20), with the question: "For each of the items, indicate the level of limitation anbout the following functions", using a 0-10 point scale, considering 0 no limitation and 10 severe limitation. Participants will rate before treatment and 24 months after treatment.
Change in masticatory rhythm at 6 months | Before treatment and 6 months after treatment
  Change in masticatory rhythm will be assessed as chewing cycle duration (in msec) measuring the the time taken to perform the 20 masticatory cycles of Optozeta's test and divided by 20. Participants will perform masticatory tests before and 6 months after treatment.
Change in masticatory rhythm at 24 months | Before treatment and 24 months after treatment
  Change in masticatory rhythm will be assessed as chewing cycle duration (in msec) measuring the the time taken to perform the 20 masticatory cycles of Optozeta's test and divided by 20. Participants will perform masticatory tests before and 24 months after treatment.
Change in masticatory laterality at 6 months | Before treatment and 6 months after treatment
  Change in masticatory laterality will be assessed by using the Asymmetry masticatory index, as = (number of right strokes - number of left strokes)/(number of right strokes + number of left strokes). Participants will perform masticatory tests before and 6 months after treatment.
Change in masticatory laterality at 24 months | Before treatment and 24 months after treatment
  Change in masticatory laterality will be assessed by using the Asymmetry masticatory index, as = (number of right strokes - number of left strokes)/(number of right strokes + number of left strokes). Participants will perform masticatory tests before and 24 months after treatment.
Change in masticatory side-switch frequency at 6 months | Before treatment and 6 months after treatment
  Change in masticatory side-switch frequency will be assessed by using the masticatory side-switch index. The number of side switches during the 20 masticatory cycles for each assay will be determined using slow playback of the video recordings of the freestyle mastication test. In the case that this switch is a change of side from left to right or right to left, a value of "1" will be assigned. If this switch consists of a change from the right or left to central or vice versa, a value of "0.5" will be assigned. If there is no change of side, the value assigned to this chewing cycle will be "0". To determine the Side Switch Index, the number of side changes will be divided by the maximum number of changes possible during these 5 assays (95). Participants will perform masticatory tests before and 6 months after treatment.
Change in masticatory side-switch frequency at 24 months | Before treatment and 24 months after treatment
  Change in masticatory side-switch frequency will be assessed by using the masticatory side-switch index. The number of side switches during the 20 masticatory cycles for each assay will be determined using slow playback of the video recordings of the freestyle mastication test. In the case that this switch is a change of side from left to right or right to left, a value of "1" will be assigned. If this switch consists of a change from the right or left to central or vice versa, a value of "0.5" will be assigned. If there is no change of side, the value assigned to this chewing cycle will be "0". To determine the Side Switch Index, the number of side changes will be divided by the maximum number of changes possible during these 5 assays (95). Participants will perform masticatory tests before and 24 months after treatment.
Change in overjet at 6 months | Before treatment and 6 months after treatment
  Change in overjet will be assessed by measuring horizontal dicrepancy on the incisal edge of maxillary and mandibular central incisors, in mm. Participants will be examined before and 6 months after treatment.
Change in overjet at 24 months | Before treatment and 24 months after treatment
  Change in overjet will be assessed by measuring horizontal dicrepancy on the incisal edge of maxillary and mandibular central incisors, in mm. Participants will be examined before and 24 months after treatment.
Change in overbite at 6 months | Before treatment and 6 months after treatment
  Change in overbite will be assessed by measuring the vertical dicrepancy on the incisal edge of maxillary and mandibular central incisors, in mm. Participants will be examined before and 6 months after treatment.
Change in overbite at 24 months | Before treatment and 24 months after treatment
  Change in overbite will be assessed by measuring the vertical dicrepancy on the incisal edge of maxillary and mandibular central incisors, in mm. Participants will be examined before and 24 months after treatment.
Change in occlusal contact area at 6 months | Before treatment and 6 months after treatment
  Change in occlusal contact area will be assessed by using interocclusal records and considering occlusal contact a distance < of 200 µm between upper and lower teeth. Occlusal records at the intercuspal position will be taken before and 6 months after treatment.
Change in occlusal contact area at 24 months | Before treatment and 24 months after treatment
  Change in occlusal contact area will be assessed by using interocclusal records and considering occlusal contact a distance < of 200 µm between upper and lower teeth. Occlusal records at the intercuspal position will be taken before and 24 months after treatment.
Change in bite force at 6 months | Before treatment and 6 months after treatment
  Change in unilateral bite force will the evaluated biting a gnathodynamometer (in Newtons). Bite force will be determined before and 6 months after treatment.
Change in bite force at 24 months | Before treatment and 24 months after treatment
  Change in unilateral bite force will the evaluated biting a gnathodynamometer (in Newtons). Bite force will be determined before and 24 months after treatment.
Change in dental mobility at 6 months | Before treatment and 6 months after treatment
  Change in dental mobility will be assessed by using the a PerioTest device. Values range from -8 (no mobility) to 50 (maximum mobility). Dental mobility will be determined before and 6 months after treatment.
Change in dental mobility at 24 months | Before treatment and 24 months after treatment
  Change in dental mobility will be assessed by using the a PerioTest device. Values range from -8 (no mobility) to 50 (maximum mobility). Dental mobility will be determined before and 24 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Willaert, DDS PhD, Study Director — University of Barcelona
Locations (1):
- Hospital Odontologic Universitat de Barcelona, L'Hospitalet de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data could be shared under a reasonable request

REFERENCES:
- [Background] Ayuso-Montero R, Mariano-Hernandez Y, Khoury-Ribas L, Rovira-Lastra B, Willaert E, Martinez-Gomis J. Reliability and Validity of T-scan and 3D Intraoral Scanning for Measuring the Occlusal Contact Area. J Prosthodont. 2020 Jan;29(1):19-25. doi: 10.1111/jopr.13096. Epub 2019 Jul 21. PMID 31270888
- [Background] Schimmel M, Christou P, Miyazaki H, Halazonetis D, Herrmann FR, Muller F. A novel colourimetric technique to assess chewing function using two-coloured specimens: Validation and application. J Dent. 2015 Aug;43(8):955-64. doi: 10.1016/j.jdent.2015.06.003. Epub 2015 Jun 22. PMID 26111925
- [Background] Riera-Punet N, Martinez-Gomis J, Willaert E, Povedano M, Peraire M. Functional limitation of the masticatory system in patients with bulbar involvement in amyotrophic lateral sclerosis. J Oral Rehabil. 2018 Mar;45(3):204-210. doi: 10.1111/joor.12597. Epub 2017 Dec 30. PMID 29240971
- [Background] Khoury-Ribas L, Ayuso-Montero R, Rovira-Lastra B, Peraire M, Martinez-Gomis J. Reliability of a new test food to assess masticatory function. Arch Oral Biol. 2018 Mar;87:1-6. doi: 10.1016/j.archoralbio.2017.12.006. Epub 2017 Dec 9. PMID 29241026
- [Background] Martinez-Gomis J, Willaert E, Nogues L, Pascual M, Somoza M, Monasterio C. Five years of sleep apnea treatment with a mandibular advancement device. Side effects and technical complications. Angle Orthod. 2010 Jan;80(1):30-6. doi: 10.2319/030309-122.1. PMID 19852636
- [Background] Uniken Venema JAM, Doff MHJ, Joffe-Sokolova DS, Wijkstra PJ, van der Hoeven JH, Stegenga B, Hoekema A. Dental side effects of long-term obstructive sleep apnea therapy: a 10-year follow-up study. Clin Oral Investig. 2020 Sep;24(9):3069-3076. doi: 10.1007/s00784-019-03175-6. Epub 2019 Dec 20. PMID 31863188